CLINICAL TRIAL: NCT02207387
Title: A Sensorimotor Contingency-based Musical Walking Program for People Living With Parkinson's Disease
Brief Title: Ambulosono Rasagiline Musical Walking Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H13-02074
Record Dates: First submitted 2014-07-28; First posted 2014-08-04 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline; Exercise; Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (5):
- MCW (Experimental): Music Contingent Walking (MCW) group: study-specific musical device that measures gait and plays music in a portable manner as the participant is walking is set at a threshold individually calculated per participant, and the music will stop playing when walking strides fall below this threshold.
  Interventions: Behavioral: Exercise; Other: Music
- NCMW (Experimental): Non-contingent Music Walking (NCMW) group: music on all the time regardless of the stride size.
  Interventions: Behavioral: Exercise; Other: Music
- NMW (Experimental): Non-music walking (NMW/silent) group: no music on at all regardless of step size.
  Interventions: Behavioral: Exercise
- MCW+rasagiline (Experimental): Music contingent walking with rasagiline group: same paradigm as the previous MCW, but with rasagiline prescribed as adjunct therapy.
  Dosage: 0.5 mg/day for the first 2 weeks to be subsequently increased to 1 mg/day
  Interventions: Drug: Azilect; Behavioral: Exercise; Other: Music
- MMW+rasagiline (Experimental): Non-music (silent) walking with rasagiline group: same paradigm as the previous NMW, but with rasagiline prescribed as adjunct therapy.
  Dosage: 0.5 mg/day for the first 2 weeks to be subsequently increased to 1 mg/day
  Interventions: Drug: Azilect; Behavioral: Exercise

INTERVENTIONS:
Drug: Azilect — Rasagiline is Parkinson's medication that can be taken alone early in the disease or with other medication and is hypothesized to produce synergistic effects with exercise.
  Other Names: rasagiline
  Arms: MCW+rasagiline; MMW+rasagiline
Behavioral: Exercise — Walking and other forms of exercise have been seen clinically and in numerous research studies to be effective against Parkinson's symptoms.
Other: Music
  Arms: MCW; MCW+rasagiline; NCMW

SUMMARY:
This study will investigate the effects of a contingency-based musical walking intervention program called Ambulosono on neural mechanisms in the brain. The investigators will investigate the long-term impact of Ambulosono on brain plasticity with functional MRI technique. Participants will undergo 3 months of Ambulosono training and their pre-training and post-training fMRI brain scans will be compared to understand the neural networks and brain mechanisms following this intervention. The investigators hypothesized that Ambulosono may induce functional compensatory reorganization of neural networks in the brain. This project will allow us to address the important potential confound of placebo influence and to aid in optimizing this intervention program. Additionally, the investigators are hoping to investigate the synergistic effects of rasagiline and exercise; the investigators' hypothesis is that there will be a positive synergistic effect, and that exercise will augment the effectiveness of rasagiline in treating Parkinson's symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Over 19 years of age
* Confirmed diagnosis of Parkinson's Disease
* Can walk 5 to 10 minutes unassisted
* Have a safe place to walk (outdoor or indoor)
* Have mild to moderate Parkinson's disease (HY1-3)
* Be able to lay flat in the scanner for the period of the study
* No reliance on wheelchair or other walking aid for ambulation
* Absence of any other serious medical conditions such as hearing impairment and dementia
* No history of other neurological and psychiatric illnesses
* No recent musculoskeletal impairment or injuries that may prevent walking

Exclusion Criteria:

* Under 19 years of age
* Unconfirmed PD diagnosis
* Require walking aid, wheelchair-bound
* No access to safe walking pathway
* Severe PD (Hoehn & Yahr stages>3)
* Impaired hearing
* Atypical Parkinsonism
* Concurrent dementia
* Recent knee, hip or foot injury (need permission from doctor)

Exclusion Criteria for fMRI

* Pacemaker
* Brain aneurysm clip
* Cochlear implant
* Recent surgery within the past 6 weeks
* Possibility of pregnancy
* Electrical stimulator for nerves or bones
* Implanted infusion pump
* History of any eye injury involving metal fragments
* History of working with metals (grinding, machining, or welding)
* Artificial heart valve
* Orthopaedic hardware (artificial joint, plate, screws, rods)
* Other metallic prostheses
* Coil, catheter or filter in any blood vessel
* Ear or eye implant
* Recent tattoos within the past 6 weeks
* Shrapnel, bullets, or other metallic fragments
* Medication releasing skin patches (nicotine, birth control, nitroglycerine)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in brain imaging signals (fMRI) | one month and four months
  resting state data task-evoked data cortical thickness volume sizes of specified brain structures

SECONDARY OUTCOMES:
Change from baseline in motor symptoms of PD | baseline and one month and four months
  Motor Symptoms:
  1. UPDRS-III scores
  2. Time taken to perform TUG and One Leg Stand Balance Test
  3. Gait performance observed from Line Walking Test, 6-Minute Walking Test, Coordinated Arm and Leg Swing Test
Change from baseline in cognition of PD | baseline and one month and four months
  Cognition:
  1. MOCA scores
  2. Changes in reaction times (Simple Reaction Time Test, Trail Making Test A and B)
  3. Performance on Phonemic Verbal Fluency Test

OTHER OUTCOMES:
Changes in mood | baseline and one month and four months
  1. Beck's Inventory for Depression
  2. Beck's Inventory for Anxiety
  3. Parkinson Fatigue Scale
Changes in impact/quality of life | baseline and one month and four months
  PDQ-39 Quality of Life Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Martin J McKeown, MD, Principal Investigator — University of British Columbia; Silke Cresswell, MD, Principal Investigator — University of British Columbia
Locations (1):
- Pacific Parkinson's Research Centre, Vancouver, British Columbia, Canada